CLINICAL TRIAL: NCT06952621
Title: A Multicenter, Randomized Controlled Clinical Study Comparing Neoadjuvant Toripalimab Combined With Nab-paclitaxel and Platinum Versus Neoadjuvant Docetaxel Combined With Cisplatin and 5-fluorouracil (DCF) in the Treatment of Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Treatment of Toripalimab Combined With Nab-paclitaxel and Platinum Versus Neoadjuvant Docetaxel Combined With Cisplatin and 5-fluorouracil (DCF) in Esophageal Squamous Cell Carcinoma
Acronym: TD-NEOE3V3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K202504-09
Record Dates: First submitted 2025-04-11; First posted 2025-05-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: toripalimab; DCF; neoadjuvant
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 cycles (Toripalimab + chemotherapy) (Experimental): Participants receive totally 3 cycles of Toripalimab combined with nab-paclitaxel and cisplatin during neoadjuvant period
  Interventions: Drug: 3 cycles (Toripalimab + chemotherapy)
- 3 cycles（DCF） (Active Comparator): Participants receive totally 3 cycles of Docetaxel combined with Cisplatin and 5-FU (5-fluorouracil) during neoadjuvant period
  Interventions: Drug: 3 cycles（DCF）

INTERVENTIONS:
Drug: 3 cycles (Toripalimab + chemotherapy) — Toripalimab: 240mg, intravenous infusion, on Day 1, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment; Nab-paclitaxel: 125mg/m², intravenous infusion, on Day 1 and Day 8, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment; Cisplatin: 75mg/m², intravenous infusion, on Day 1, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment;
  Arms: 3 cycles (Toripalimab + chemotherapy)
Drug: 3 cycles（DCF） — Docetaxel: 70mg/m², intravenous infusion, on day 1, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment; Cisplatin: 70mg/m², intravenous infusion, on day 1, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment; 5-FU (5-fluorouracil): 750mg/m², intravenous infusion, on day 1 to day 5, every 3 weeks (Q3W), for 3 cycles of neoadjuvant treatment
  Arms: 3 cycles（DCF）

SUMMARY:
This study is a randomized, controlled, open-label, multicenter Phase III clinical trial, designed to evaluate the efficacy and safety of neoadjuvant toripalimab in combination with nab-paclitaxel and platinum versus neoadjuvant docetaxel in combination with cisplatin and 5-fluorouracil (DCF) in the treatment of resectable locally advanced esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria are eligible to participate in the study:

  1. Voluntarily sign the written informed consent form;
  2. Age 18-75 years, inclusive of 18 and 75 years, both male and female;
  3. Life expectancy of ≥3 months;
  4. Expected to achieve R0 resection;
  5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
  6. Patients with resectable locally advanced (T1 N1-3 M0 or T2-4a N0-3 M0 (T2≥3cm or poorly differentiated)) thoracic esophageal squamous cell carcinoma confirmed by histology and who have not previously received treatment;
  7. No suspicious metastatic lymph nodes in the neck (excluding regional lymph nodes in the upper thoracic esophageal cancer area) as suggested by neck ultrasound or enhanced CT, and no systemic metastasis detected by imaging studies;
  8. Presence of a definite tumor lesion;
  9. Good organ function as indicated by screening laboratory test results:

     1. Hematology (no blood transfusions or treatment with blood products or granulocyte colony-stimulating factor within 14 days): Neutrophil count (NEU) ≥1.5×10⁹/L (1,500/mm³); Platelet (PLT) count ≥100×10⁹/L (100,000/mm³); Hemoglobin ≥90 g/L.
     2. Liver: Total bilirubin (TBil) ≤1.5×ULN; or for participants with total bilirubin levels <1.5×ULN, direct bilirubin within normal limits; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN;
     3. Kidney: Serum creatinine ≤1.5×ULN or calculated creatinine clearance (CrCl) ≥60 mL/min (using the Cockcroft-Gault formula);
     4. Coagulation function: International normalized ratio (INR) ≤1.5, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤1.5×ULN;
  10. Fertile males or females of childbearing potential must use effective contraception methods (such as oral contraceptives, intrauterine devices, or barrier methods combined with spermicides) during the trial and continue contraception for 6 months after the end of treatment;
  11. Good compliance and willingness to cooperate with follow-up visits.

Exclusion Criteria:

* Patients who meet any of the following criteria are ineligible for this study:

  1. Previous treatment with PD-1/PD-L1 agents or drugs targeting another T-cell receptor (e.g., CTLA-4, OX-40, etc.);
  2. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
  3. Active autoimmune disease or suspicion of such, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc., with the exception of type 1 diabetes and hypothyroidism controlled with stable-dose replacement therapy, and skin diseases not requiring systemic treatment (e.g., psoriasis, vitiligo);
  4. History of interstitial lung disease ≥ Grade 2;
  5. Received systemic corticosteroids (prednisone >10mg/day or equivalent) or other immunosuppressive drugs within 14 days prior to the first study drug administration;
  6. History of immunodeficiency, including other acquired or congenital immunodeficiency diseases, history of organ transplantation, or having undergone allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
  7. Received live vaccine within 4 weeks prior to the first study drug administration;
  8. Presence of severe cardiovascular and cerebrovascular diseases:

     1. Uncontrolled hypertension or pulmonary arterial hypertension;
     2. Unstable angina or myocardial infarction, coronary artery bypass grafting, or stent implantation within 6 months prior to study drug administration;
     3. Chronic heart failure with cardiac function ≥ Grade 2 (New York Heart Association [NYHA] classification);
     4. Left ventricular ejection fraction (LVEF) <50%;
     5. Severe arrhythmias requiring drug treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia). For example: male QTcF >450 msec or female QTcF >470 msec, complete left bundle branch block, third-degree atrioventricular block;
     6. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to study drug administration;
  9. Presence of uncontrollable or severe underlying diseases, including but not limited to active infections requiring systemic antibiotic therapy;
  10. Positive test results for human immunodeficiency virus (HIV) antibodies, active hepatitis B or C. The following cases are allowed to participate in this study:

      1. Positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg), but HBV DNA below the detection limit of the study center (negative) or <500IU/ML, and after clinical treatment and presentation, the investigator determines that there is no active infection;
      2. Positive for hepatitis C antibody, but HCV RNA below the detection limit of the study center (negative);
  11. Known active tuberculosis (TB). Patients suspected of having active TB must be excluded by chest X-ray, sputum tests, and clinical symptoms and signs;
  12. Presence of other active malignancies within the past 2 years, excluding malignancies that are expected to be cured after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell carcinoma of the skin, or ductal carcinoma in situ of the breast treated with radical surgery);
  13. History of substance abuse or mental disorders that cannot be controlled;
  14. Pregnant or breastfeeding women;
  15. Presence of other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities that, in the investigator's judgment, may increase the risk associated with participation in the study or may interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | Pathological detection after surgery within 1 month

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | Pathological detection after surgery within 1 month
objective response rate (ORR) | From enrollment to the period before surgery (4-6 weeks after the third cycle of treatment).
event-free survival (EFS) | from randomization to disease progression that makes surgery impossible, postoperative disease progression, local or distant recurrence, or death from any cause (whichever occurs first，assessed up to 60 months)
overall survival | from randomization to death from any cause，assessed up to 60 months
Adverse events | form date of enrollment until the end of the study, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospitial, Xi'an, Shaanxi Rrovince, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No